CLINICAL TRIAL: NCT05821192
Title: A Prospective Clinical Study of Chemotherapy Plus Programmed Death-1 Monoclonal Antibody in the Treatment of Refractory or Relapsed Peripheral T Cell Lymphoma Not Otherwise Specified and Angioimmunoblastic T-cell Lymphoma.
Brief Title: Chemotherapy Plus PD-1 Monoclonal Antibody in the Treatment of Refractory or Relapsed Peripheral T-cell Lymphoma.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ou Bai, MD/PHD (Other)
Collaborators: Second Hospital of Jilin University (Other); China-Japan Union Hospital, Jilin University (Other)
Responsible Party: Sponsor-Investigator, Ou Bai, MD/PHD, Professor, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rrPTCL-R-PD1-001
Record Dates: First submitted 2023-03-23; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Peripheral T-Cell Lymphoma, Not Otherwise Specified; Angioimmunoblastic T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell; Immunoblastic Lymphadenopathy | interventions — Rituximab; Gemcitabine; Dexamethasone; Cisplatin; spartalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R-GDP plus PD-1 monoclonal antibody (Experimental): Rituximab, Gemcitabine, Cisplatin, Dexamethasone, PD-1 monoclonal antibody
  Interventions: Drug: Rituximab; Drug: Gemcitabine; Drug: Dexamethasone; Drug: Cisplatin; Drug: PD-1 monoclonal antibody

INTERVENTIONS:
Drug: Rituximab — 375mg/m2 by IV infusion once every 3 weeks
Drug: Gemcitabine — 1 g/m2 on Days 1 by IV infusion once every 3 weeks
Drug: Dexamethasone — 40 mg on Days 1 to 4 of each 3-week cycle by IV infusion
Drug: Cisplatin — 75 mg/m2 on Days 1 by IV infusion once every 3 weeks
Drug: PD-1 monoclonal antibody — 200mg on Days 2 by IV infusion once every 3 weeks

SUMMARY:
A multi-center, prospective clinical study to evaluate the efficacy and safety of R-GDP plus PD-1 monoclonal antibody in the treatment of refractory or relapsed peripheral T cell lymphoma not otherwise specified and Angioimmunoblastic T-cell lymphoma, which has previously shown promising efficacy.

DETAILED DESCRIPTION:
Objective to evaluate the efficacy and safety of R-GDP (Rituximab, Gemcitabine, Dexamethasone, Cisplatin) plus PD-1 monoclonal antibody in patients with refractory or relapsed peripheral T cell lymphoma not otherwise specified or Angioimmunoblastic T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with peripheral T cell lymphoma not otherwise specified or Angioimmunoblastic T-cell lymphoma confirmed by histopathology;
2. Age 18 to 70 years for all sexs;
3. Progressive disease or no response in patients who have received first-line chemotherapy (at least 2 cycles), and patients who refuse or can't suffer from intravenous chemotherapy;
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
5. Life expectancy ≥ 3 months;
6. There are measurable lesions (lymph nodes enlargement, nodal masses, enlargement of lymphoid organs and extranodal lesion that are measurable in two diameters (longest diameter and shortest diameter). A measurable node must have an longest diameter greater than 1.5 cm. A measurable extranodal lesion should have an longest diameter greater than 1.0 cm.);
7. Function of organs:

   1. Hepatic function: Total bilirubin ≤ 1.5 times upper limit of normal (ULN), direct bilirubin ≤ 1.5 times ULN; aspartate aminotransferase (AST) or Alanine aminotransferase （ALT） ≤ 2.5 times ULN (5 times ULN if liver involvement with lymphoma);
   2. Bone marrow function (without growth factor in 7 days before the first drugs): WBC ≥ 2.0×109/l; ANC ≥ 1.0×109/l; PLT ≥ 50×109/l; Hb ≥ 8g/dl;
   3. Renal function: Creatinine ≤ 1.5 times ULN or creatinine clearance rate ≥ 30ml/min or creatinine clearance rate ≤ 2.5 times ULN;
   4. Pulmonary function: blood oxygen saturation ≥ 95% in resting state without oxygen inhalation;
   5. Coagulation function: international normalised ratio (INR) ≤ 1.5 times ULN and activated partial thromboplastin time (aPTT) ≤ 1.5 times ULN (Patients whose prolonged PT or increased INR resulted in clotting factor inhibitors, should be selected at the investigator's discretion);
   6. Heart function: LVEF ≥ 50%;

Exclusion Criteria:

1. Unrelieved toxic reaction CTCAE grade > 1 before the first drugs in this research (except adverse effects that won't affect this study, estimated by the investigator, such as alopecia);
2. There is an active infection, including but not limited to known active tuberculosis, known latent tuberculosis, herpes zoster and pneumonia;
3. Patient is known to be positive for Human immunodeficiency virus (HIV) infection; Or serological status reflect active hepatitis B virus(HBV) infection or active hepatitis C virus (HCV) infection:

   1. Patients with HBsAg(+), HBcAb (+) or HBsAg (+) should detect HBV-DNA. Patients who has HBV-DNA ≤ 1000IU/ml and agree to have anti-HBV therapy can be selected;
   2. Patients with HCVAb (+) and HCV RNA < 15 IU/mL can be selected;
4. Heart failure with New York Heart Association （NYHA） grade III or IV, unstable angina pectoris, severe ventricular arrhythmias with poor control, acute myocardial ischemia showed by electrocardiogram or had myocardial infarction in 6 months before screening. Or patients can't suffer from chemotherapy due to other heart function disorders, estimated by investigator;
5. Intractable nausea or vomiting that can't be controlled by supportive care, chronic gastrointestinal diseases or dysphagia of capsules, or had intestinal resection which may affect the drug absorption;
6. The investigator determined or other evidence showed patients have severe or poorly controlled systemic diseases, including poorly controlled hypertension and active bleeding body constitution. Patients with thrombotic diseases such as pulmonary embolism and deep venous thrombosis are also not suitable to participate in this study;
7. Patients have interstitial pneumonia or once had chemotherapy-induced interstitial pneumonia during chemotherapy, who have treatment risk in the estimation of investigator;
8. Pregnant or lactating women;
9. The investigator determine the patients having other infectors which may affect compliance;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2023-04-18 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 16 months
  Percentage of Complete remission (CR), and Partial remission (PR).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 24 months
  Progression-free survival#PFS# is defined as the time from the date of enrollment to the date of first documentation of progressive disease (PD) or death from any cause.
Overall survival (OS) | 24 months
  Overall survival#OS# is defined as the time from the date of enrollment to the date of death from any cause.
Incidence of adverse events (AEs) | 24 months
  Any untoward medical occurrence in a clinical investigational participant administered a medicinal product which does not necessarily have a causal relationship with this treatment.
Serious Adverse Event (SAE) | 24 months
  A serious adverse event will be considered any undesirable sign, symptom, or medical condition with one or more of the following outcomes:
  1. is fatal, is life-threatening
  2. requires or prolongs inpatient hospitalization
  3. results in persistent or significant disability/incapacity
  4. constitutes a congenital anomaly or birth defect

CONTACTS AND LOCATIONS:
Overall Officials: Ou Bai, doctor, Study Chair — The First Hospital of Jilin University
Locations (1):
- The First Bethune Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No